CLINICAL TRIAL: NCT05760742
Title: Evaluation of the Protective Effects of a Novel Dietary Microalgae Supplement (PeLiv) Following Exercise-induced Muscle Damage and Influence on Endurance Capacity After Prolonged Consumption
Brief Title: Evaluation of the Effects of a Novel Dietary Microalgae Based Ingredient on Muscle Recovery and Endurance Capacity
Acronym: PORPHY-ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microphyt (Industry)
Collaborators: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00004940
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: recovery; muscle endurance; exercise capacity; microalgae; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator): 2 capsules of Maltodextrin per day
  Interventions: Dietary Supplement: Placebo
- MicAlgae100 (Experimental): 2 capsules per day containing 100mg of microalgae based ingredient
  Interventions: Dietary Supplement: MicAlgae
- MicAlgae250 (Experimental): 2 capsules per day containing 250mg of microalgae based ingredient
  Interventions: Dietary Supplement: MicAlgae
- MicAlgae500 (Experimental): 2 capsules per day containing 500mg of microalgae based ingredient
  Interventions: Dietary Supplement: MicAlgae

INTERVENTIONS:
Dietary Supplement: MicAlgae — 2 months of supplementation with an innovative microalgae based ingredient
  Arms: MicAlgae100; MicAlgae250; MicAlgae500
Dietary Supplement: Placebo — 2 months of supplementation with a placebo (Maltodextrin)
  Arms: Placebo group

SUMMARY:
The purpose of this investigation is to examine the effects of consuming a new dietary microalgae based supplement vs. placebo on neuromuscular function, energy utilization, soreness, perceptual wellness, swelling, and markers of muscle damage and inflammation in healthy young men before and after an acute exercise-induced muscle damage protocol (downhill running), and influence on endurance capacity after prolonged consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* Healthy as assessed by Medical and activity history questionnaire (MHQ)
* Recreationally active according to American College of Sports Medicine guidelines
* Able to provide written and dated informed consent to participate in the study

Exclusion Criteria:

* Untrained
* Any response of "yes" on the PAR-Q+
* Physical limitations preventing running, countermovement jump, and strength (peak isometric torque and peak isokinetic torque) assessments

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Neuromuscular function | From 0 to week 4
  isokinetic peak torque in Newton per meter (N/m)

SECONDARY OUTCOMES:
Energy utilization (Oxygen consumption - VO2) | From 0 to week 4
  Running economy during a 5-minute run at 80% of the speed at VO2max with gaz exchange analyzis
Energy utilization (Oxygen consumption - VO2) | From 0 to week 8
  Running economy during a 5-minute run at 80% of the speed at VO2max with gaz exchange analyzis
Isokinetic neuromuscular function | From 0 to week 8
  peak torque in Newton per meter (N/m)
Isometric neuromuscular function | From 0 to week 8
  peak torque in Newton per meter (N/m)
Endurance capacity | From 0 to week 4
  Maximal oxygen consumption (VO2max) determined during graded exercise test
Endurance capacity | From 0 to week 8
  Maximal oxygen consumption (VO2max) determined during graded exercise test
Soreness and perceptual wellness | From 0 to week 4
  Evaluated using using a 100-point numerical pain rating scale anchored with 0= no pain to 100= the most intense pain sensation imaginable after exercise-induced muscle damage protocol
Soreness and perceptual wellness | From 0 to week 8
  Evaluated using using a 100-point numerical pain rating scale anchored with 0= no pain to 100= the most intense pain sensation imaginable after exercise-induced muscle damage protocol
Swelling - Muscle thickness (mm or cm) | From 0 to week 4
  Evaluated using musculoskeletal ultrasound
Swelling - overall thigh circumference (mm or cm) | From 0 to week 4
  Evaluated using musculoskeletal ultrasound
Creatine kinase (UI/I) | After 4 weeks of supplementation
  Blood marker analyzis
lactate dehydrogenase (U/L) | After 4 weeks of supplementation
  Blood marker analyzis
Myoglobin (ug/l) | After 4 weeks of supplementation
  Blood marker analyzis
Interleukin-6 (pg/ml) | After 4 weeks of supplementation
  Blood marker analyzis - inflammation
Tumor necrosis factor-α (ug/ml) | After 4 weeks of supplementation
  Blood marker analyzis - inflammation
C-reactive protein (mg/l) | After 4 weeks of supplementation
  Blood marker analyzis - inflammation
Isometric Neuromuscular function | From 0 to week 4
  Peak torque in Newton per meter (N/m)

CONTACTS AND LOCATIONS:
Overall Officials: David Fukuda, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No